CLINICAL TRIAL: NCT00329615
Title: Insulin Treatment in Cancer Cachexia: Effects on Survival, Metabolism and Physical Functioning. A Randomized Prospective Study.
Brief Title: Insulin Treatment in Cancer Cachexia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Swedish Cancer Foundation (Other); Medical Research Council (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: kl450112
Record Dates: First submitted 2006-05-23; First posted 2006-05-25 (Estimated); Last update posted 2009-08-21 (Estimated); Status verified 2009-08

CONDITIONS: Cancer Cachexia
Keywords: Cancer cachexia; Tumor host metabolism
MeSH Terms: interventions — Isophane Insulin, Human

INTERVENTIONS:
Drug: Insulatard, flexpen

SUMMARY:
The study is designed to evaluate whether daily insulin treatment to weight losing cancer patients attenuates progression of cancer cachexia and improves metabolism.

DETAILED DESCRIPTION:
Randomized study with long-term follow-up based on survival, health related quality of life, food intake, resting energy expenditure, body composition, exercise capacity and measurement of metabolic efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Weight loss
* Systemic solid cancer

Exclusion Criteria:

* Diabetes
* Brain metastases
* Expectant survival of less than 6 months
* Serum creatinine above 200 umol/l
* Persistent of recurrent fever
* Cholestasis

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135
Dates: Start 2000-01; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Health related quality of life,
food intake,
resting energy expenditure,
body composition,
metabolic efficiency,
spontaneous physical activity,
blood and hormonal tests
serum tumor markers

SECONDARY OUTCOMES:
Survival

CONTACTS AND LOCATIONS:
Overall Officials: Kent G Lundholm, MD, Principal Investigator — Department of Surgery, Göteborg University
Locations (1):
- Department of Surgery, Inst of Clinical Sciences, Gothenburg, Sweden

REFERENCES:
- [Derived] Wallengren O, Bosaeus I, Lundholm K. Dietary energy density, inflammation and energy balance in palliative care cancer patients. Clin Nutr. 2013 Feb;32(1):88-92. doi: 10.1016/j.clnu.2012.05.023. Epub 2012 Jun 23. PMID 22727547